CLINICAL TRIAL: NCT06438562
Title: Evaluation of Vitamin A Absorption From Fortified Bouillon Using Post-prandial Retinyl Ester Response in Comparison With an Oil-based Vitamin A Supplement
Brief Title: Evaluation of Vitamin A Absorption From Fortified Bouillon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Particles for Humanity, PBC (Industry); Tropical Diseases Research Centre, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-0327; A074600 (Other: UW- Madison); CALS/NUTRITIONAL SCIENCES (Other: UW- Madison); Version 10/2/2024 (Other: UW- Madison)
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Vitamin A
MeSH Terms: interventions — Vitamin A; Oils

STUDY DESIGN:
Intervention Model Description: Participants will receive all 3 study treatments over 3 treatment periods.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized and blinded to all treatments and treatment sequence.
  Care providers and investigators are blinded to experimental treatments and treatment sequence.
  Outcome assessors are blinded to all treatments and treatment sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin A #1 (Experimental): Bouillon fortified with vitamin A formulation #1 plus unfortified oil
  Interventions: Other: Bouillon fortified with vitamin A #1 plus unfortified oil
- Vitamin A #2 (Experimental): Bouillon fortified with vitamin A formulation #2 plus unfortified oil
  Interventions: Other: Bouillon fortified with vitamin A #2 plus unfortified oil
- Unfortified bouillon positive control (Active Comparator): Unfortified bouillon plus vitamin A fortified oil
  Interventions: Other: Unfortified bouillon plus vitamin A in oil

INTERVENTIONS:
Other: Unfortified bouillon plus vitamin A in oil — Participants consume unfortified bouillon with vitamin A oil
  Arms: Unfortified bouillon positive control
Other: Bouillon fortified with vitamin A #1 plus unfortified oil — Participants consume vitamin A #1 fortified bouillon plus unfortified oil
  Arms: Vitamin A #1
Other: Bouillon fortified with vitamin A #2 plus unfortified oil — Participants consume vitamin A #2 fortified bouillon plus unfortified oil
  Arms: Vitamin A #2

SUMMARY:
The goal of this clinical trial is to measure how well different formulations of vitamin A (VA) are absorbed by the body when they are added to bouillon (broth) as vitamin A palmitate (VAP). Fortifying bouillon cubes with VA is one potential approach to addressing VA deficiency, which is a major public health issue in many low- and lower-income countries. The main question this study aims to answer is to compare the amount of VA that is absorbed by the body from three different VAP formulations that are added to bouillon.

Participants will consume different formulations of VA and have multiple blood collections.

DETAILED DESCRIPTION:
This study is being conducted to help characterize the absorption of 3 different formulations of VAP (PFH-VAP and BASF-VAP250 vs a positive control) when prepared as broth with an oil dose containing VAP or placebo (referred to as the "study treatments") and consumed by healthy adult women of reproductive age (ages 18 - 49 years).

Participants will undergo 3 treatment periods and will be blinded to treatment sequence using a 3-period, 3-treatment crossover design to receive all 3 treatments. All 3 treatment periods will include blood sampling to measure VA levels from pre- through 24 hours post-broth consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonpregnant women
* ≥18 and <49 years of age
* Able and willing to provide informed consent
* Body mass index (BMI) between 18.5 to 30.0 kg/m2
* Willing and able to undergo study procedures, including: repeated blood sampling, a baseline hemoglobin and pregnancy test, adherence to a low-vitamin A diet at specified times throughout the study, consumption of provided meals (specifically, a breakfast of bouillon, peanut butter, and a bagel or bread), and, except for the Screening visit, foregoing alcohol for at least 2 days before each visit and fasting for ≥8 hours before each visit

Exclusion Criteria:

* Currently pregnant
* Breastfeeding a child under 1 year of age
* Allergic to soy or peanut butter
* Current use of smoking tobacco products or any other form of nicotine
* Active eating disorder diagnosis
* Current diagnosis of acute or chronic illness, including hepatitis, Celiac's disease, Crohn's disease, and cystic fibrosis
* Moderate or severe anemia according to World Health Organization guidelines (i.e., hemoglobin ≤10.9 g/dL)
* Unable or unwilling to refrain from consuming alcohol when required
* Unable or unwilling to discontinue consumption of foods that are high in vitamin A and of vitamin A supplements when required during the study
* Taking prescription oral medication that includes a retinoid, e.g., isotretinoin/ Accutane
* Taking proton pump inhibitors.
* Unable/unwilling to avoid taking antacids during the fasting period prior to sample collection
* Unable/unwilling to fast for periods of at least 10 hours at a time
* Status relationship with a member of the study team.
* Unable to fulfill study requirements per the judgment of the investigator

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Serum retinyl ester area-under-the-effect-curve | Baseline to 8 hours
  The serum retinyl ester area-under-the-effect-curve (corrected for baseline retinyl ester concentrations) will be calculated for each treatment to determine relative absorption of vitamin A, (nmol/L*h)
Serum retinyl ester area-under-the-effect-curve | Baseline to 24 hours
  The serum retinyl ester area-under-the-effect-curve (corrected for baseline retinyl ester concentrations) will be calculated for each treatment to determine relative absorption of vitamin A, (nmol/L*h)

SECONDARY OUTCOMES:
Serum retinol maximum concentration (Cmax) | Baseline to 24 hours
  Maximum serum retinol concentration observed, (µmol/L)
Serum retinyl ester maximum concentration (Cmax) | Baseline to 24 hours
  Maximum serum retinyl ester concentration observed, (nmol/L)
Time to maximum serum retinol concentration (Tmax) | Baseline to 24 hours
  Time to maximum serum retinol concentration, (h)
Time to serum retinyl ester maximum concentration (Tmax) | Baseline to 24 hours
  Time to maximum serum retinyl ester concentration, (h)

OTHER OUTCOMES:
Total body vitamin A using retinol isotope dilution | Baseline
  The retinol isotope dilution test provides an estimate of total body stores of vitamin A, (umol)
Liver vitamin A concentrations using retinol isotope dilution | Baseline
  The retinol isotope dilution test provides an estimate of liver vitamin A concentrations, (umol/g)
C-reactive protein | Baseline
  To determine inflammation at each treatment visit, (mg/L)
Serum carotenoids | Baseline
  Serum carotenoid concentrations will be measured using high-performance liquid chromatography at baseline for each treatment visit, (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Tanumihardjo, PhD, Principal Investigator — University of Wisconsin, Madison; Bryan M Gannon, PhD, Study Director — University of Wisconsin, Madison; Luke M Funk, MD, MPH, Study Director — University of Wisconsin, Madison; Justin Chileshe, PhD, Study Director — Tropical Diseases Research Centre, Zambia
Locations (2):
- University of Wisconsin-Madison, Madison, Wisconsin, United States
- Tropical Diseases Research Centre - Field Office, Rufunsa, Zambia

IPD SHARING:
Plan to Share IPD: No